CLINICAL TRIAL: NCT04586439
Title: A Randomized, Open-Label, Parallel, Single Dose Study to Investigate Pharmacokinetics, Safety, and Tolerability of JNJ-73763989 in Healthy Chinese Adult Participants
Brief Title: A Study of JNJ-73763989 in Healthy Chinese Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108867; 73763989HPB1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Panel A: JNJ-73763989 (Experimental): Participants will receive single subcutaneous (SC) injection of low dose of JNJ-73763989 on Day 1.
  Interventions: Drug: JNJ-73763989
- Panel B: J NJ-73763989 (Experimental): Participants will receive single SC injection of high dose of JNJ-73763989 on Day 1.
  Interventions: Drug: JNJ-73763989

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 will be administered (high or low dose) as single SC injection.

SUMMARY:
The purpose of the study is to evaluate the single-dose Pharmacokinetics of JNJ-73763976 and JNJ-73763924 following a subcutaneous (SC) injection of JNJ-73763989 (JNJ-3989) in healthy Chinese adult participants at 2 different doses, Dose 1 (Panel A) or Dose 2 (Panel B).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy based on physical examination, laboratory assessment, vital signs and electrocardiogram (ECG) at screening
* A female participant of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [hCG]) pregnancy test at screening and a negative urine pregnancy test on Day -1
* A male participant must agree not to donate sperm after enrollment (Day 1) in the study and a female participant must agree not to donate eggs (ova, oocytes) during the study until at least 90 days after receiving the study drug
* Participant must not use nicotine-containing substances including tobacco products for at least 3 months prior to screening until completion of the study
* Participant must have suitable veins for cannulation and/or repeated venipuncture

Exclusion Criteria:

* Participant with a history of cardiac arrhythmias (example, premature ventricular contractions), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Participant with human immunodeficiency virus infection (confirmed by antibodies) at screening
* Participant with current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B infection (confirmed by HBsAg), or hepatitis C virus (HCV) infection (confirmed by HCV antibody), or hepatitis E infection (confirmed by hepatitis E antibody IgM) at screening
* Participant has positive test result(s) for alcohol and/or drugs of abuse (including amphetamines, benzodiazepines, cocaine, cannabinoids, opioids, and methadone) at screening and Day-1
* Participant has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit, or confound the protocol-specified assessments. This may include but is not limited to renal dysfunction estimated Glomerular Filtration Rate (GFR) <60 millimeter per minute (mL/min) /1.73 m^2 at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 4 Weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Plasma Concentration of JNJ-73763989 | Predose up to 48 hours postdose (up to Day 3)
  Plasma samples will be analyzed to determine concentrations of JNJ-73763989 (as the 2 triggers JNJ-73763976 and JNJ-73763924).
Urine Concentration of JNJ-73763989 | Predose up to 48 hours postdose (up to Day 3)
  Urine samples will be analyzed to determine concentrations of JNJ-73763989 (as the 2 triggers JNJ-73763976 and JNJ-73763924).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Li H, Niu X, Zhang Y, Zhang D, Zhang Y, Wang L, Miao Y, Jiang Y, Ji J, Chen Q, Wu X, Ediage EN, Kakuda TN, Biermer M. Pharmacokinetics, Safety, and Tolerability of the siRNA JNJ-73763989 in Healthy Chinese Adult Participants. Clin Pharmacol Drug Dev. 2023 Feb;12(2):175-180. doi: 10.1002/cpdd.1197. Epub 2022 Nov 22. PMID 36415122